CLINICAL TRIAL: NCT05589311
Title: Transformative Learning to Virtual Inter-Professional Education in Musculoskeletal Pain: A Randomised Trial
Brief Title: Transformative Learning to Virtual Inter-Professional Education in Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022/2048
Record Dates: First submitted 2022-03-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Pain
Keywords: Pain education; Healthcare professionals; Interprofessional education; Transformative Learning
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): One-time 2.5-hour virtual lecture on musculoskeletal pain conducted following Transformative Learning principles
  Interventions: Other: Transformative Learning principles
- Control group (Active Comparator): One-time 2.5-hour virtual lecture on musculoskeletal pain conducted using conventional didactic approach
  Interventions: Other: Conventional didactic approach

INTERVENTIONS:
Other: Transformative Learning principles — Transformative Learning principles are incorporated into the pain education workshop to stimulate critical reflection and critical discourse during the learning process.
  Arms: Intervention group
Other: Conventional didactic approach — The conventional didactic approach focuses on lecture-based instruction as the teaching center, emphasizing the delivery of syllabus and concept.
  Arms: Control group

SUMMARY:
Musculoskeletal (MSK) pain is amongst the leading reasons for people seeking medical attention in local primary care, accounting for 6-28% of principal diagnoses. Patient education is one of the important treatment strategies to ease pain, reduce suffering and disability. However, from our anecdotal experience, patients often report there is an inconsistency in the information being provided by healthcare professionals. This can be due to the existence of different MSK pain frameworks as the understanding of pain sciences evolves. Hence, there is a need for regular Continuous Medical Education (CME) to update and improve healthcare staff knowledge and skills on this aspect in Singapore.

The conventional teaching method is typically used in SingHealth Polyclinics (SHP) CME sessions. It focuses on lecture-based instruction as the teaching centre, emphasizing the delivery of syllabus and concept. The conventional teaching method has been shown to be less effective than other teaching strategies (e.g. Case based learning) in practical application and critical thinking abilities. Mezirow proposed the use of Transformative Learning to enhance adult learning. We aim to conduct an RCT to investigate whether this teaching method is superior to the conventional teaching method in improving MSK pain knowledge, management advice, attitudes and beliefs of healthcare professionals in primary care.

This randomised multi-centre, prospective study will be conducted across all SHP polyclinics. Healthcare professionals working in SHP will be invited to participate in the study. Participants in both the intervention and control groups will be asked to complete the questionnaires at 3 time-points: before and after the lecture, as well as 1 month later. The anonymised data collected will then be analysed using descriptive and inferential statistics.

DETAILED DESCRIPTION:
Study Design

This randomised, multi-centre, prospective study will be conducted in all public primary care centres also known as polyclinics which manage patients with acute and chronic medical conditions. Patients may also visit the polyclinics which are located mainly in the eastern, southern and north-eastern part of Singapore, to utilise the vaccination, medical examination or screening, and/ or allied health services such as physiotherapy and podiatry services.

This project will seek approval from the institutional ethics committee prior to commencement and it will be conducted in accordance with the Declaration of Helsinki.

Participants

SHP conducts regular continuing education lectures as part of the ongoing effort in ensuring continual development of knowledge and skills of the healthcare workforce. These lectures provide opportunity for staff to achieve professional self-improvement and to ensure that their knowledge and skills are up-to-date and relevant.

The MSK pain lectures will be incorporated as one of continuing education sessions. The delivery of the MSK pain lecture will be scheduled to be conducted online. Invitation email will be sent to healthcare professionals. Information about the lecture and study will be stated in the email (sample attached). Those who are interested in the lecture and agree to participate in the study will register interest by providing their email address. The lecture Zoom link will be sent to the participants before the lecture commencement.

The participants who are involved in the study will be anonymised i.e. their personal identifications will not be collected during the study.

The lecture invitation email will state that an education research will be conducted to evaluate and compare the effectiveness of two Zoom training methods. And that the participants will be randomized into either one of the methods. Data collection form link will be sent to them. As the study is completely voluntary, it is possible that the participants can sign up for the lecture but choose not to attempt the questionnaire forms or participate in the study at any time-point. The data collection is anonymous, hence it is impossible to identify the participants who do not fill up the questionnaires.

Randomization

Participants will be randomized in a 1:1 ratio to either intervention or control group according to a computer generated block randomization list. Random permuted blocks are used to ensure balance over time. The block size is determined by the statistician and will kept confidential from the study team until final database lock. Each participant will be assigned a study ID and the intervention/control assignment. Intervention and control group will receive the email links respectively to the virtual lectures.

Sample size

Based on the study by Collearya et al., to detect a significant increase in scores for Management Advice Vignette between the groups (increase in score of 25 in intervention group and increase in score of 3 in control group for the question on Exercise), the minimum required sample size for individual (block) randomization is 47 per arm, with a power of 80% and 5% significance level.

Virtual Lecture

A 2.5-hour virtual lecture will be conducted online. Pain science, common MSK conditions and management in primary care, basic pharmacology in pain management and pain education will be covered during the lecture. The educational materials will be developed using various pain resources such as relevant sections in the textbook by Wall and Melzack, patients' and clinicians' guidebooks of explaining pain by Butler and Moseley, and other related healthcare literatures such as clinical practice guidelines and systematic reviews of MSK conditions. The educational slides provide no specific explanations about the individual items in the evaluation tools such as NPQ, CAV, MAV and HC-PAIRS.

Intervention group: Lecture conducted using Transformative Learning principles. Control group: Lecture conducted using conventional didactic approach with Q&A session after the slides presentation.

Both groups will receive the same content but provided using different education conceptual framework.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals working in SingHealth Polyclinics

Exclusion Criteria:

* Healthcare professionals working in institutions other than SingHealth Polyclinics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Learner's reactions and reflection form (LRRF) | after the intervention (lecture)
  This self-developed evaluation form was developed to gather participants' feedback on the lecture and the learning experience. Participants are required to answer 18 questions using a 1 to 10 scale where 1 is strongly disagree and 10 is strongly agree.
Change in Neurophysiology of Pain Questionnaire (NPQ) | Up to 1 month pre-intervention, immediate post-intervention (lecture) and 1 month follow up
  NPQ will be used to evaluate the participants' understanding of pain neurophysiology. It is a 12-item validated questionnaire. Each item has three response options: true, false, undecided. The NPQ uses the number-correct scoring method, whereby the total number of correct answers is added to create an overall score. 1 point is awarded for each correct response. A score of 0 is attributed to incorrect responses and those marked as undecided.
  Comparison of pre-intervention and post-intervention (immediate and 1 month follow up) NPQ scores (assessed through number of correct answers).
Change in Clinical Assessment Vignette (CAV) | Up to 1 month pre-intervention, immediate post-intervention (lecture) and 1 month follow up
  6 Common MSK conditions Assessment Questions, modified from Moroz (2017). It is a quiz to test the knowledge of the participants on the common MSK conditions. A short description is provided on the patient's signs and symptoms and the participant is required to identify the correct diagnosis.
  Comparison of pre-intervention and post-intervention (immediate and 1 month follow up) CAV scores (assessed through number of correct answers).
Change in Health care Pain Attitudes and Impairment Relationship Scale (HC-PAIRS) | Up to 1 month pre-intervention, immediate post-intervention (lecture) and 1 month follow up
  HC-PAIRS is derived by altering Pain and Impairment Relationship scale (PAIRS) developed by Riley et al. Items are scored by the location of responses on the Likert scales following each question, with items 1, 6, and 14 scored by reversing the numbers. Items 10 and 13 were omitted from the original version, as recommended by Houben et al., to improve the construct of the scale. Scores of individual items are totalled, yielding the HC-PAIRS score.
  Comparison of pre-intervention and post-intervention (immediate and 1 month follow up) HC-PAIRS scores (assessed on a 7-point Likert scale).
Change in Management Advice Vignette (MAV) | Up to 1 month pre-intervention, immediate post-intervention (lecture) and 1 month follow up
  4 MSK Management Advice Questions (Bishop et al. 2008). It is a quiz to assess the appropriateness of MSK pain management recommendations of the participants. A clinical case vignette is provided and the participant is required to answer short multiple choice questions regarding the appropriate management advice. It is an indirect measure of the clinical behaviour.
  Comparison of pre-intervention and post-intervention (immediate and 1 month follow up) MAV scores (assessed through number of correct answers).

CONTACTS AND LOCATIONS:
Overall Officials: Khim Siong Ng, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colleary G, O'Sullivan K, Griffin D, Ryan CG, Martin DJ. Effect of pain neurophysiology education on physiotherapy students' understanding of chronic pain, clinical recommendations and attitudes towards people with chronic pain: a randomised controlled trial. Physiotherapy. 2017 Dec;103(4):423-429. doi: 10.1016/j.physio.2017.01.006. Epub 2017 Mar 22. PMID 28797666
- [Background] Moseley L. Unraveling the barriers to reconceptualization of the problem in chronic pain: the actual and perceived ability of patients and health professionals to understand the neurophysiology. J Pain. 2003 May;4(4):184-9. doi: 10.1016/s1526-5900(03)00488-7. PMID 14622702
- [Background] Catley MJ, O'Connell NE, Moseley GL. How good is the neurophysiology of pain questionnaire? A Rasch analysis of psychometric properties. J Pain. 2013 Aug;14(8):818-27. doi: 10.1016/j.jpain.2013.02.008. Epub 2013 May 4. PMID 23651882
- [Background] Moroz A. Clinical Reasoning Workshop: Lumbosacral Spine and Hip Disorders. MedEdPORTAL. 2017 Sep 20;13:10632. doi: 10.15766/mep_2374-8265.10632. PMID 30800833
- [Background] Riley JF, Ahern DK, Follick MJ. Chronic pain and functional impairment: assessing beliefs about their relationship. Arch Phys Med Rehabil. 1988 Aug;69(8):579-82. PMID 3408327
- [Background] Rainville J, Bagnall D, Phalen L. Health care providers' attitudes and beliefs about functional impairments and chronic back pain. Clin J Pain. 1995 Dec;11(4):287-95. doi: 10.1097/00002508-199512000-00006. PMID 8788576
- [Background] Houben RM, Vlaeyen JW, Peters M, Ostelo RW, Wolters PM, Stomp-van den Berg SG. Health care providers' attitudes and beliefs towards common low back pain: factor structure and psychometric properties of the HC-PAIRS. Clin J Pain. 2004 Jan-Feb;20(1):37-44. doi: 10.1097/00002508-200401000-00008. PMID 14668655
- [Background] Bishop A, Foster NE, Thomas E, Hay EM. How does the self-reported clinical management of patients with low back pain relate to the attitudes and beliefs of health care practitioners? A survey of UK general practitioners and physiotherapists. Pain. 2008 Mar;135(1-2):187-95. doi: 10.1016/j.pain.2007.11.010. PMID 18206309
- [Background] Keyte D, Richardson C. Re-thinking pain educational strategies: Pain a new model using e-learning and PBL. Nurse Educ Today. 2011 Feb;31(2):117-21. doi: 10.1016/j.nedt.2010.05.001. Epub 2010 Jun 20. PMID 20566232
- [Derived] Ng KS, Tang ZY, Wong PNF, Chua JLJ, Goh LLL, Koh YLE, Koh KH. Integrating transformative learning theory in synchronous E-learning in musculoskeletal pain education among primary care nurses: a randomized study. BMC Nurs. 2025 Jul 7;24(1):858. doi: 10.1186/s12912-025-03540-9. PMID 40624538